CLINICAL TRIAL: NCT04969185
Title: Associations Between Drug Levels and the Risk of Malaria and Drug Resistance in the Setting of Seasonal Malaria Chemoprevention in Bobo-Dioulasso, Burkina Faso
Brief Title: Association Between Drug Levels, Malaria, and Antimalarial Resistance in the Setting of Seasonal Malaria Chemoprevention
Acronym: DRUMARS
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21-33890
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Malaria,Falciparum
Keywords: seasonal malaria chemoprevention; sulfadoxine-pyrimethamine; amodiaquine; antimalarial resistance; pharmacokinetics; falciparum malaria; malnutrition
MeSH Terms: conditions — Malaria, Falciparum; Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be used to determine: (1) the levels of exposure to SDX, PYR, and AQ; (2) presence of malaria parasitemia; and (3) characterize markers of antimalarial drug resistance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Children eligible to receive SMC diagnosed with uncomplicated Plasmodium falciparum malaria: Children eligible to receive SMC (6-59 months of age) who were diagnosed with uncomplicated P. falciparum malaria at the health facility.
- Group 2: Children eligible to receive SMC presenting at health facility without malaria parasitemia: Group 2 will be defined as children eligible to receive SMC (6-59 months of age) who presented at the health facility and tested negative for malaria parasitemia.This group will serve as the control group to Group 1 Cases to compare the SP-AQ drug levels between children who did and did not get malaria.
- Group 3: Children 5-10 years of age diagnosed with uncomplicated Plasmodium falciparum malaria: Group 3 will be defined as children ineligible to receive SMC (5-10 years of age) who were diagnosed with uncomplicated P. falciparum malaria at the health facility. This group will serve as the control group to Group 1 Cases to compare the prevalence of SP and AQ resistance markers.

SUMMARY:
In areas of the Sahel sub-region of Africa with intense seasonal malaria transmission, seasonal malaria chemoprevention (SMC) with sulfadoxine-pyrimethamine and amodiaquine (SP+AQ) has become the standard-of-care for the prevention of malaria in children. Despite the scale-up of SMC across West Africa, the malaria burden remains high. Reasons for this are not well understood, however, it is hypothesized that children eligible for SMC who get malaria may be underdosed or may have not received SP+AQ. Moreover, there are major concerns that the continued use of the SMC strategy may increase selection of AQ and/or SP-resistant Plasmodium falciparum parasites. The overall objective of this observational study are to understand the factors driving malaria among children eligible to receive SMC and whether circulating levels of sulfadoxine (SDX), pyrimethamine (PYR), and AQ are associated with risks of malaria and antimalarial drug resistance.

DETAILED DESCRIPTION:
In areas of the Sahel sub-region of Africa with intense seasonal malaria transmission, seasonal malaria chemoprevention (SMC) with sulfadoxine-pyrimethamine and amodiaquine (SP+AQ) has become the standard-of-care for the prevention of malaria in children. Despite the scale-up of SMC across West Africa, the malaria burden remains high. Reasons for this are not well understood, however, it is hypothesized that children eligible for SMC who get malaria may be underdosed or may have not received SP+AQ. Moreover, there are major concerns that the continued use of the SMC strategy may increase selection of AQ and/or SP-resistant Plasmodium falciparum parasites. The overall objective of this observational study are to understand the factors driving malaria among children eligible to receive SMC and whether circulating levels of sulfadoxine (SDX), pyrimethamine (PYR), and AQ are associated with risks of malaria and antimalarial drug resistance. The specific objectives of this study are as follows:

1. To determine associations between the levels of exposure to the components of SP+AQ (SDX, PYR, and AQ) and malaria risk.
2. To determine associations between levels of exposure to the components of SP+AQ and the prevalence of P. falciparum genetic polymorphisms associated with drug resistance.
3. To compare the prevalence of genetic polymorphisms associated with SP+AQ resistance between parasites infecting children eligible to receive SMC and those infecting older children ineligible to receive SMC.
4. To assess whether the prevalence of genetic polymorphisms associated with SP+AQ resistance changes over time.

ELIGIBILITY:
The inclusion criteria will differ for each group enrolled into the study:

Inclusion criteria for Group 1 (Children 6-59 months of age diagnosed with uncomplicated P. falciparum malaria):

* Aged 6-59 months
* Resident of health facility catchment area
* Provision of parental consent
* Fever (temperature of ≥37.5°C) or history of fever in the past 24 hours
* Confirmed P. falciparum parasitemia by RDT and/or microscopy

Inclusion criteria for Group 2 (Children 6-59 months of age without malaria):

* Aged 6-59 months
* Resident of health facility catchment area
* Provision of parental consent
* Negative for P. falciparum parasitemia by RDT and/or microscopy

Inclusion criteria for Group 3 (Children 5-10 years of age diagnosed with uncomplicated P. falciparum malaria):

* Aged 5-10 years
* Resident of health facility catchment area
* Provision of parental consent
* Fever (temperature of ≥37.5°C) or history of fever in the past 24 hours
* Confirmed P. falciparum parasitemia by RDT and/or microscopy

The exclusion criteria for all children are as follows:

* Refusal to participate
* Residence outside of health facility catchment areas
* Known treatment of malaria (not SMC) in the past 14 days
* Danger signs (lethargy, unable to drink or breast feed, repeated vomiting, unable to stand or sit due to weakness)
* Signs of severe malaria, including altered conscious, respiratory distress (rapid breathing), severe anemia (<5 g/dL), or other signs of organ dysfunction.
* Non-malarial illness that is severe or prevents necessary study procedures

Ages: 6 Months to 10 Years | Sex: All
Age Groups: Child
Study Population: The target population will be children residing in the catchment areas of study health facilities within Bobo-Dioulasso, Burkina Faso.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Risk of parasitemia | during the seasonal SMC campaign period over three years
  Detected by blood smear microscopy
Prevalence of antimalarial resistance markers associated with SP | during the seasonal SMC campaign period over three years
  Prevalence of pfdhfr and pfdhps mutations
Prevalence of antimalarial resistance markers associated with AQ | during the seasonal SMC campaign period over three years
  Prevalence of pfcrt and pfmdr1 mutations

CONTACTS AND LOCATIONS:
Overall Officials: Philip Rosenthal, MD, Principal Investigator — University of California, San Francisco; Jean-Bosco Ouédraogo, MD PhD, Principal Investigator — Institut de Recherche en Sciences de la Santé, Burkina Faso
Locations (2):
- Burkina Faso (2):
  - Colsama Health Facility, Bobo-Dioulasso
  - Sakaby Health Facility, Bobo-Dioulasso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roh ME, Zongo I, Haro A, Huang L, Some AF, Yerbanga RS, Conrad MD, Wallender E, Legac J, Aweeka F, Ouedraogo JB, Rosenthal PJ. Seasonal Malaria Chemoprevention Drug Levels and Drug Resistance Markers in Children With or Without Malaria in Burkina Faso: A Case-Control Study. J Infect Dis. 2023 Oct 3;228(7):926-935. doi: 10.1093/infdis/jiad172. PMID 37221018